CLINICAL TRIAL: NCT04069091
Title: Implementation of Prevention and Intervention of Maternal Perinatal Depression to Strengthen Maternal and Child Health
Acronym: IMPRINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Katri Räikkönen (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Katri Räikkönen, Professor of Psychology, University of Helsinki
Organization: University of Helsinki (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Perinatal Depression

STUDY DESIGN:
Intervention Model Description: Please note, that November 1 2024, the study design was changed to a single-arm clinical trial; previous a two-arm cluster-randomized clinical trial.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT intervention (Experimental): Participants in the CBT intervention arm will undergo standard antenatal care and the 'Enjoy your Bump' (iloodottaa.fi) online self-help intervention employing elements of cognitive behavioral therapy (CBT)
  Interventions: Behavioral: 'Enjoy your Bump' (iloodottaa.fi) online self-help intervention
- Standard care (No Intervention): Participants in the Standard Care arm will undergo standard antenatal care.

INTERVENTIONS:
Behavioral: 'Enjoy your Bump' (iloodottaa.fi) online self-help intervention — The intervention employs elements of cognitive behavioral therapy: empathic, clear and sensitive communication with women and their families, problem self-formulation of solutions to problems, behavioral activation, identification and changing negative automated negative thoughts, addressing low confidence, and promoting problem- solving and relapse prevention.
  The Enjoy your Bump intervention has been adapted to the Finnish culture and healthcare setting (ilodottaa.fi).
  Arms: CBT intervention

SUMMARY:
IMPRINT strengthens maternal and child health by screening, treating and preventing maternal perinatal depression, the most common complication of pregnancy and the child's first 1000 days. It is associated with poor pregnancy outcome and perinatal mortality and has adverse consequences on physical and mental development of the child. Yet, only 7-28% of women with perinatal depression worldwide receive appropriate evidence-based care. This is astounding given that the need of investing on mental health is widely recognized and low-intensity interventions not requiring costly mental health professionals have been shown to be effective.

IMPRINT improves the effectiveness, reliability, safety, appropriateness, equity and efficiency of routine health care provided for the mother and the child during the child's first 1000 days of life. The investigators 1) have adapted into the gender-, country-, and cultural-context an existing evidence-based, low-intensity pregnancy intervention targeting maternal perinatal depression (online CBT-based therapy) (iloodottaa.fi); 2) test in cluster-randomised trial the short- and long-term efficacy of the intervention in women who report clinically relevant, subthreshold or more severe symptoms in an early pregnancy depression screen; 3) study biological, psychological and social determinants of depressive symptom severity, comorbidities and response to interventions. The study recruits women from 58 antenetal clinics in the cities of Helsinki, Vantaa, Keski-Uusimaa, Kuopio and Lohja and aims at recruiting 500 women to the intervention and 500 women to the control arms.

Because of low recruitment rate, the cluster-randomized clinical trial design was changed to a single-arm clinical trial. All pregnant mothers who meet the inclusion criteria are eligible to participate in the CBT-intervention. In parallel with the change in study design, recruitment expanded to cover all antenatal clinical in the well-being services counties: Helsinki, Vantaa and Kerava, Central Uusimaa, Western Uusimaa (Lohja), Eastern Finland, and Pirkanmaa. Amendment to HUS ethical committee, approval date: June 26 2024; Amendment to HUS research permit, approval date: August 8 2024; Approvals from the counties participating in the study, approval dates: by October 31 2024.

ELIGIBILITY:
Inclusion Criteria:

* EPDS screen result of 10 or more
* Agreed to be invited for the intervention during the screening phase

Exclusion Criteria:

* Active suicidality
* Presence of severe mental disorder
* Concurrent use of psychotropic medication / concurrently under psychosocial treatment for mental disorder

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | Measured immediately after intervention at 26-28 gestational weeks
  The primary outcome in the women is depressive symptoms measured using the Edinburgh Postnatal Depression Scale (EPDS). The EPDS is a self-report questionnaire consisting of a single scale of 10 items, each rated 0-3. Higher total scores (range 0-30) indicate more depressive symptomatology, and scores of at least 10 indicate clinically relevant depressive symptoms, i.e. probable depression.
Child developmental milestones | Measured at 3 months of corrected age after childbirth
  The primary outcome in the children is child developmental milestones measured using the Ages and Stages-3 questionnaires (ASQ-3). The ASQ-3 comprises 30 age-appropriate items measuring communication, gross motor, fine motor, problem solving and personal/social skills. Each domain comprises six questions with response 'yes' (scored 10) indicating the child can master the skill, 'sometimes' (scored 5) if the skill is emerging or occasional, and 'not yet' (scored 0) if the child is not able perform the skill. Highest domain scores (range 0-60) indicate mastery of the skill. On each domain, scores over 2 standard deviations (SD) below the mean for the age indicate developmental delay, scores between 1-2 SDs below the mean indicate mild developmental delay, and scores higher than one SD below the mean indicate typical development.

CONTACTS AND LOCATIONS:
Overall Officials: Katri Räikkönen, PhD, Principal Investigator — University of Helsinki
Locations (1):
- University of Helsinki, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No